CLINICAL TRIAL: NCT00380874
Title: A Randomized, Double-Blind, Placebo-Controlled Trial Of The Prevention And Treatment Of Chemotherapy-Induced Peripheral Neuropathy Symptoms In Subjects With Advanced Colorectal Cancer
Brief Title: Prevention And Treatment Of Chemotherapy-Induced Peripheral Neuropathy In Subjects With Advanced Colorectal Cancer
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See detailed description for termination reason
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081124
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Results first posted 2009-04-17 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2009-10

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy
Keywords: Pain; chemotherapy
MeSH Terms: conditions — Pain | interventions — Pregabalin; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): flexible dosing
  Interventions: Drug: Pregabalin
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — 150- 600 mg/day (double blind in divided doses)
  Other Names: Chemotherapy
  Arms: 1
Drug: Placebo — Placebo
  Other Names: Chemotherapy
  Arms: 2

SUMMARY:
Prevention and treatment of the severity of symptoms of chemotherapy-induced peripheral neuropathy.

DETAILED DESCRIPTION:
This study was terminated on July 15, 2008. The results of an interim analysis showed that the conditional power to detect a difference in treatment groups was insufficient to warrant study continuation and therefore termination of the trial was recommended. The decision to terminate the trial was not based on safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cytological confirmed carcinoma of the Colon Stage III (Dukes C) or metastatic Colorectal Cancer (Dukes D)
* Independent of this protocol, the patient has decided to receive standard of care for the treatment of cancer with oxaliplatin combined with 5-fluorouracil/folinic acid (5-FU/FA) for a minimum of 9 cycles

Exclusion Criteria:

* Presence of neuropathic pain or peripheral polyneuropathy or identified causes of painful paresthesia including radiotherapy-induced or malignant plexopathy, lumbar or cervical radiculopathy existing prior to baseline
* Any patients who are not suitable to be treated with either Oxaliplatin and/or 5-FU/FA or pregabalin according to the respective local labeling

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- Australia (2):
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, Adelaide, South Australia
- Germany (3):
  - Pfizer Investigational Site, Bielefeld
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Hamm
- Italy (2):
  - Pfizer Investigational Site, Chieti Scalo
  - Pfizer Investigational Site, Potenza
- South Korea (2):
  - Pfizer Investigational Site, Goyang-si, Gyeonggi-do
  - Pfizer Investigational Site, Seoul
- Spain (3):
  - Pfizer Investigational Site, Santander, Cantabria
  - Pfizer Investigational Site, Alicante
  - Pfizer Investigational Site, Jaén
- Taiwan (2):
  - Pfizer Investigational Site, Niao-Sung Hsiang, Kaohsiung Hsien
  - Pfizer Investigational Site, Taipei

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081124&StudyName=Prevention%20And%20Treatment%20Of%20Chemotherapy-Induced%20Peripheral%20Neuropathy%20Symptoms%20In%20Subjects%20With%20Adv.%20Colorectal%20Cancer.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 69 subjects screened, 64 were randomized, and 61 received treatment. Of the 8 subjects screened but not treated, 1 was ineligible due to an abnormal laboratory test result, 6 were ineligible due to a reason categorized as other, and 1 was no longer willing to continue in the study.
Groups:
- Pregabalin: Pregabalin 150 to 600 milligrams per day (mg/day) flexible dose + chemotherapy (oxaliplatin combined with 5-fluorouracil/folinic acid (5-FU/FA). Possible dose levels of pregabalin were 150 mg/day (75 mg capsules twice a day [BID]), 300 mg/day (150 mg capsules BID) or 600 mg/day (300 mg capsules BID).
- Placebo: matching placebo + chemotherapy (oxaliplatin combined with 5-fluorouracil/folinic acid (5-FU/FA).
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 32 | 29
Completed | 19 | 19
Not Completed | 13 | 10
Not completed — Adverse Event | 7 | 7
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Not related to study drug | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 32 | 29 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (11.3) | 56.1 (12.9) | 57.6 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 21 | 21 | 42

OUTCOME MEASURES:

1. Secondary Outcome: Duration Adjusted Average Change (DAAC) of Paresthesic Symptom Score Within Each Cycle of Chemotherapy Measured by Numeric Rating Scale (NRS)
Description: Least squares mean of change: mean at cycle minus mean at Baseline. Paresthetic Duration Adjusted Average Change (DAAC) endpoint was computed based on Numeric Rating Scale (NRS) of paresthesia (collected 0=no pain; 1-3=mild pain; 4-6=moderate pain; 7-10=severe pain). DAAC endpoint is defined as the Area Under Curve (AUC) of the collected NRS over time, divided by collection time period (up to 10 days).
Time Frame: Baseline to Cycle 9
Population: Intent-to-Treat (ITT) population: subjects with at least 1 dose of study medication and for whom at least 1 post-baseline efficacy evaluation was obtained.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 32 | 29
score on scale
  Cycle 1 (n=25, 27) | 0.03 (0.06) | 0.13 (0.05)
  Cycle 2 (n=26, 26) | 0.35 (0.16) | 0.22 (0.16)
  Cycle 3 (n=24, 23) | 0.53 (0.21) | 0.37 (0.21)
  Cycle 4 (n=25, 23) | 0.64 (0.21) | 0.40 (0.22)
  Cycle 5 (n=24, 22) | 1.03 (0.33) | 0.53 (0.35)
  Cycle 6 (n=21, 21) | 0.74 (0.28) | 0.64 (0.28)
  Cycle 7 (n=17, 22) | 0.93 (0.30) | 0.96 (0.26)
  Cycle 8 (n=16, 19) | 0.83 (0.29) | 1.03 (0.27)
  Cycle 9 (n=16, 18) | 0.92 (0.36) | 1.65 (0.34)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Cycle 1. Sample size was based on original primary efficacy parameter (PEP) of time to persistent paresthesia symptoms (symptoms developing in 35% of subjects taking pregabalin and 60% taking placebo symptoms). Assuming Type I error rate of 0.05 and a 2-sided log-rank test for equality of time to persistent symptoms survival curves, the study would have had at least 90% power using 100 subjects per treatment group. The original PEP was modified to secondary due to lack of symptom emergence; Test type: Superiority or Other; p = 0.2536, ANCOVA — Cycle 1. No multiple comparisons adjustment was made; Model terms include treatment, study center, and baseline score; Mean Difference (Final Values) = -0.09, Standard Error of Mean 0.08 — LS means and corresponding standard errors derived from ANCOVA model were used
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Cycle 2. Sample size was based on original primary efficacy parameter (PEP) of time to persistent paresthesia symptoms (symptoms developing in 35% of subjects taking pregabalin and 60% taking placebo symptoms). Assuming Type I error rate of 0.05 and a 2-sided log-rank test for equality of time to persistent symptoms survival curves, the study would have had at least 90% power using 100 subjects per treatment group. The original PEP was modified to secondary due to lack of symptom emergence; Test type: Superiority or Other; p = 0.5757, ANCOVA — No multiple comparisons adjustment was made; Model terms include treatment, study center, and baseline score; Mean Difference (Final Values) = 0.13, Standard Error of Mean 0.23 — LS means and corresponding standard errors derived from ANCOVA model were used
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Cycle 3. Sample size was based on original primary efficacy parameter (PEP) of time to persistent paresthesia symptoms (symptoms developing in 35% of subjects taking pregabalin and 60% taking placebo symptoms). Assuming Type I error rate of 0.05 and a 2-sided log-rank test for equality of time to persistent symptoms survival curves, the study would have had at least 90% power using 100 subjects per treatment group. The original PEP was modified to secondary due to lack of symptom emergence; Test type: Superiority or Other; p = 0.6065, ANCOVA — No multiple comparisons adjustment was made; Model terms include treatment, study center, and baseline score; Mean Difference (Final Values) = 0.15, Standard Error of Mean 0.30 — LS means and corresponding standard errors derived from ANCOVA model were used
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Cycle 4. Sample size was based on original primary efficacy parameter (PEP) of time to persistent paresthesia symptoms (symptoms developing in 35% of subjects taking pregabalin and 60% taking placebo symptoms). Assuming Type I error rate of 0.05 and a 2-sided log-rank test for equality of time to persistent symptoms survival curves, the study would have had at least 90% power using 100 subjects per treatment group. The original PEP was modified to secondary due to lack of symptom emergence; Test type: Superiority or Other; p = 0.4301, ANCOVA — No multiple comparisons adjustment was made; Model terms include treatment, study center, and baseline score; Mean Difference (Final Values) = 0.24, Standard Error of Mean 0.31 — LS means and corresponding standard errors derived from ANCOVA model were used
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Cycle 5. Sample size was based on original primary efficacy parameter (PEP) of time to persistent paresthesia symptoms (symptoms developing in 35% of subjects taking pregabalin and 60% taking placebo symptoms). Assuming Type I error rate of 0.05 and a 2-sided log-rank test for equality of time to persistent symptoms survival curves, the study would have had at least 90% power using 100 subjects per treatment group. The original PEP was modified to secondary due to lack of symptom emergence; Test type: Superiority or Other; p = 0.3125, ANCOVA — No multiple comparisons adjustment was made; Model terms include treatment, study center, and baseline score; Mean Difference (Final Values) = 0.50, Standard Error of Mean 0.49 — LS means and corresponding standard errors derived from ANCOVA model were used
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Cycle 6.Sample size was based on original primary efficacy parameter (PEP) of time to persistent paresthesia symptoms (symptoms developing in 35% of subjects taking pregabalin and 60% taking placebo symptoms). Assuming Type I error rate of 0.05 and a 2-sided log-rank test for equality of time to persistent symptoms survival curves, the study would have had at least 90% power using 100 subjects per treatment group. The original PEP was modified to secondary due to lack of symptom emergence; Test type: Superiority or Other; p = 0.8169, ANCOVA — No multiple comparisons adjustment was made; Model terms include treatment, study center, and baseline score; Mean Difference (Final Values) = 0.09, Standard Error of Mean 0.41 — LS means and corresponding standard errors derived from ANCOVA model were used
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Cycle 7. Sample size was based on original primary efficacy parameter (PEP) of time to persistent paresthesia symptoms (symptoms developing in 35% of subjects taking pregabalin and 60% taking placebo symptoms). Assuming Type I error rate of 0.05 and a 2-sided log-rank test for equality of time to persistent symptoms survival curves, the study would have had at least 90% power using 100 subjects per treatment group. The original PEP was modified to secondary due to lack of symptom emergence; Test type: Superiority or Other; p = 0.9359, ANCOVA; Model terms include treatment, study center, and baseline score; Mean Difference (Final Values) = -0.03, Standard Error of Mean 0.40 — LS means and corresponding standard errors derived from ANCOVA model were used
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Cycle 8. Sample size was based on original primary efficacy parameter (PEP) of time to persistent paresthesia symptoms (symptoms developing in 35% of subjects taking pregabalin and 60% taking placebo symptoms). Assuming Type I error rate of 0.05 and a 2-sided log-rank test for equality of time to persistent symptoms survival curves, the study would have had at least 90% power using 100 subjects per treatment group. The original PEP was modified to secondary due to lack of symptom emergence; Test type: Superiority or Other; p = 0.6233, ANCOVA; Model terms include treatment, study center, and baseline score; Mean Difference (Final Values) = -0.20, Standard Error of Mean 0.40 — LS means and corresponding standard errors derived from ANCOVA model were used
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Cycle 9.Sample size was based on original primary efficacy parameter (PEP) of time to persistent paresthesia symptoms (symptoms developing in 35% of subjects taking pregabalin and 60% taking placebo symptoms). Assuming Type I error rate of 0.05 and a 2-sided log-rank test for equality of time to persistent symptoms survival curves, the study would have had at least 90% power using 100 subjects per treatment group. The original PEP was modified to secondary due to lack of symptom emergence; Test type: Superiority or Other; p = 0.1569, ANCOVA — No multiple comparisons adjustment was made; Model terms include treatment, study center, and baseline score; Mean Difference (Final Values) = -0.73, Standard Error of Mean 0.50 — LS means and corresponding standard errors derived from ANCOVA model were used

2. Secondary Outcome: Duration Adjusted Average Change (DAAC) of Dysesthesia Symptom Score Within Each Cycle of Chemotherapy Measured by Numeric Rating Scale (NRS)
Description: Least squares (LS) mean of change: mean at cycle minus mean at Baseline. Dysesthesic Duration Adjusted Average Change (DAAC) endpoint was computed based on Numeric Rating Scale (NRS) of dysesthesis (collected 0=no pain; 1-3=mild pain; 4-6=moderate pain; 7-10=severe pain). DAAC endpoint was defined as the Area Under Curve (AUC) of the collected NRS over time, divided by collection time period (up to 10 days).
Time Frame: Baseline to Cycle 9, LOCF cycle endpoint
Population: ITT population, subjects with at lest 1 dose of study medication and for whom at least 1 post-baseline efficacy evaluation was obtained.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 32 | 29
score on scale
  Cycle 1 (n=25,27) | 0.09 (0.08) | 0.13 (0.07)
  Cycle 2 (n=26,26) | 0.75 (0.25) | 0.38 (0.25)
  Cycle 3 (n=24,23) | 0.91 (0.33) | 0.65 (0.34)
  Cycle 4 (n=25,23) | 1.01 (0.37) | 0.71 (0.39)
  Cycle 5 (n=24,22) | 1.54 (0.48) | 0.80 (0.50)
  Cycle 6 (n=21,21) | 0.88 (0.38) | 0.93 (0.38)
  Cycle 7 (n=17,22) | 1.17 (0.39) | 1.17 (0.34)
  Cycle 8 (n=16,19) | 1.33 (0.40) | 1.06 (0.36)
  Cycle 9 (n=16, 18) | 1.24 (0.44) | 1.75 (0.42)
  LOCF endpoint (n=26, 27) | 1.36 (0.38) | 1.33 (0.38)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Cycle 1; Test type: Superiority or Other; p = 0.7207, ANCOVA — Model terms include treatment, study center, and baseline score; Cycle 1. No multiple comparisons adjustment was made; Mean Difference (Final Values) = -0.04, 95% CI [-0.25 to 0.17], Standard Error of Mean 0.11 — LS means and corresponding standard errors derived from ANCOVA model were used
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Cycle 2; Test type: Superiority or Other; p = 0.3111, ANCOVA — No multiple comparisons adjustment was made; Model terms include treatment, study center, and baseline score; Mean Difference (Final Values) = 0.37, 95% CI [-0.36 to 1.10], Standard Error of Mean 0.36 — LS means and corresponding standard errors derived from ANCOVA model were used
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Cycle 3; Test type: Superiority or Other; p = 0.5925, ANCOVA — No multiple comparisons adjustment was made; Model terms include treatment, study center, and baseline score; Mean Difference (Final Values) = 0.26, 95% CI [-0.70 to 1.22], Standard Error of Mean 0.48 — LS means and corresponding standard errors derived from ANCOVA model were used
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Cycle 4; Test type: Superiority or Other; p = 0.5812, ANCOVA — No multiple comparisons adjustment was made; Model terms include treatment, study center, and baseline score; Mean Difference (Final Values) = 0.30, 95% CI [-0.80 to 1.41], Standard Error of Mean 0.55 — LS means and corresponding standard errors derived from ANCOVA model were used
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Cycle 5; Test type: Superiority or Other; p = 0.2925, ANCOVA — No multiple comparisons adjustment was made; Model terms include treatment, study center, and baseline score; Mean Difference (Final Values) = 0.75, 95% CI [-0.67 to 2.16], Standard Error of Mean 0.70 — LS means and corresponding standard errors derived from ANCOVA model were used
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Cycle 6; Test type: Superiority or Other; p = 0.9276, ANCOVA — No multiple comparisons adjustment was made; Model terms include treatment, study center, and baseline score; Mean Difference (Final Values) = -0.05, 95% CI [-1.15 to 1.05], Standard Error of Mean 0.54 — LS means and corresponding standard errors derived from ANCOVA model were used
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Cycle 7; Test type: Superiority or Other; p = 0.9952, ANCOVA; Model terms include treatment, study center, and baseline score; Mean Difference (Final Values) = 0.00, 95% CI [-1.06 to 1.07], Standard Error of Mean 0.53
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Cycle 8; Test type: Superiority or Other; p = 0.6265, ANCOVA; Model terms include treatment, study center, and baseline score; Mean Difference (Final Values) = 0.27, 95% CI [-0.85 to 1.38], Standard Error of Mean 0.55 — LS means and corresponding standard errors derived from ANCOVA model were used
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Cycle 9; Test type: Superiority or Other; p = 0.4209, ANCOVA — No multiple comparisons adjustment was made; Model terms include treatment, study center, and baseline score; Mean Difference (Final Values) = -0.51, 95% CI [-1.77 to 0.76], Standard Error of Mean 0.62 — LS means and corresponding standard errors derived from ANCOVA model were used
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Last Observation Carried Forward (LOCF)endpoint; Test type: Superiority or Other; p = 0.9657, ANCOVA — No multiple comparisons adjustment was made; Model terms include treatment, study center, and baseline score; Mean Difference (Final Values) = 0.02, 95% CI [-1.06 to 1.11], Standard Error of Mean 0.54 — LS means and corresponding standard errors derived from ANCOVA model were used

3. Secondary Outcome: Duration Adjusted Average Change (DAAC) of Pain Symptom Score Within Each Cycle of Chemotherapy Measured by Numeric Rating Scale (NRS)
Description: Least squares (LS) mean of change: mean at cycle minus mean at Baseline. Pain Duration Adjusted Average Change (DAAC) endpoint was computed based on Numeric Rating Scale (NRS) of pain (collected 0=no pain; 1-3=mild pain; 4-6=moderate pain; 7-10=severe pain). DAAC endpoint was defined as the Area Under Curve (AUC) of the collected NRS over time, divided by collection time period (up to 10 days).
Time Frame: Baseline to Cycle 9, LOCF cycle endpoint
Population: ITT population: subjects with at least 1 dose of study medication and for whom at least 1 post-baseline efficacy evaluation was obtained.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 32 | 29
score on scale
  Cycle 1 (n=25,27) | 0.02 (0.06) | 0.07 (0.06)
  Cycle 2 (n=25,26) | 0.29 (0.15) | 0.16 (0.15)
  Cycle 3 (n=23,23) | 0.47 (0.24) | 0.26 (0.24)
  Cycle 4 (n=25,23) | 0.62 (0.28) | 0.27 (0.29)
  Cycle 5 (n=24,22) | 0.85 (0.33) | 0.31 (0.35)
  Cycle 6 (n=21,21) | 0.54 (0.27) | 0.58 (0.27)
  Cycle 7 (17,22) | 0.92 (0.31) | 0.60 (0.27)
  Cycle 8 (n=16,19) | 0.92 (0.36) | 0.60 (0.33)
  Cycle 9 (n=16, 18) | 0.86 (0.41) | 0.97 (0.39)
  LOCF endpoint (n=26, 27) | 0.65 (0.27) | 0.78 (0.27)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Cycle 1; Test type: Superiority or Other; p = 0.5392, ANCOVA; Mean Difference (Final Values) = -0.06, 95% CI [-0.24 to 0.12], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Cycle 2; Test type: Superiority or Other; p = 0.5412, ANCOVA; Mean Difference (Final Values) = 0.13, 95% CI [-0.30 to 0.57], Standard Error of Mean 0.22
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Cycle 3; Test type: Superiority or Other; p = 0.5358, ANCOVA; Mean Difference (Final Values) = 0.21, 95% CI [-0.48 to 0.90], Standard Error of Mean 0.34
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Cycle 4; Test type: Superiority or Other; p = 0.4059, ANCOVA; Mean Difference (Final Values) = 0.34, 95% CI [-0.48 to 1.17], Standard Error of Mean 0.41
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Cycle 5; Test type: Superiority or Other; p = 0.2712, ANCOVA; Mean Difference (Final Values) = 0.54, 95% CI [-0.44 to 1.52], Standard Error of Mean 0.49
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Cycle 6; Test type: Superiority or Other; p = 0.9181, ANCOVA; Mean Difference (Final Values) = -0.04, 95% CI [-0.81 to 0.73], Standard Error of Mean 0.38
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Cycle 7; Test type: Superiority or Other; p = 0.4357, ANCOVA; Mean Difference (Final Values) = 0.33, 95% CI [-0.52 to 1.17], Standard Error of Mean 0.42
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.5103, ANCOVA; Mean Difference (Final Values) = 0.33, 95% CI [-0.67 to 1.33], Standard Error of Mean 0.49
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Cycle 9; Test type: Superiority or Other; p = 0.8499, ANCOVA; Mean Difference (Final Values) = -0.11, 95% CI [-1.29 to 1.07], Standard Error of Mean 0.58
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; LOCF endpoint; Test type: Superiority or Other; p = 0.7359, ANCOVA; Mean Difference (Final Values) = -0.13, 95% CI [-0.90 to 0.64], Standard Error of Mean 0.39

4. Secondary Outcome: Change in Pain Scores Rated on Neuropathic Pain Symptom Inventory (NPSI) Subscales From Baseline Cycle
Description: Least squares (LS) mean of change: mean at cycle minus mean at Baseline. Neuropathic Pain Symptom Inventory (NPSI) = questionnaire designed to evaluate symptoms of neuropathic pain. 11-point numeric rating scale, range: 0 (no pain) to 10 (worst pain imaginable) best describing their average pain for last 24 hours.
Time Frame: Baseline to Cycle 9, Last Observation Carried Forward (LOCF) cycle endpoint
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 32 | 29
score on scale
  Burning spontaneous pain Cycle 3 (n=27,27) | 0.09 (0.06) | -0.02 (0.06)
  Burning spontaneous pain Cycle 4 (n=28,23) | 0.02 (0.09) | 0.15 (0.10)
  Burning spontaneous pain Cycle 5 (n=26,24) | 0.06 (0.08) | 0.19 (0.08)
  Burning spontaneous pain Cycle 6 (n=24,24) | 0.28 (0.12) | 0.14 (0.12)
  Burning spontaneous pain Cycle 7 (n=21,23) | 0.42 (0.25) | 0.40 (0.24)
  Burning spontaneous pain Cycle 8 (n=19,21) | 0.53 (0.22) | 0.23 (0.21)
  Burning spontaneous pain Cycle 9 (n=19,20) | 0.54 (0.28) | 0.59 (0.27)
  Burning spontaneous pain LOCF endpoint (n=29,27) | 0.33 (0.18) | 0.35 (019)
  Pressing spontaneous pain Cycle 2 (n=28,27) | -0.01 (0.04) | 0.05 (0.04)
  Pressing spontaneous pain Cycle 3 (n=28,24) | 0.05 (0.03) | 0.01 (0.03)
  Pressing spontaneous pain Cycle 4 (n=28,23) | 0.03 (0.08) | 0.20 (0.09)
  Pressing spontaneous pain Cycle 5 (n=26,24) | 0.06 (0.04) | 0.06 (0.04)
  Pressing spontaneous pain Cycle 6 (n=24,24) | 0.09 (0.05) | 0.09 (0.05)
  Pressing spontaneous pain Cycle 7 (n=32,29) | 0.26 (0.18) | 0.30 (0.17)
  Pressing spontaneous pain Cycle 8 (n=19,21) | 0.39 (0.15) | 0.12 (0.15)
  Pressing spontaneous pain Cycle 9 (n=19,20 | 0.25 (0.09) | 0.14 (0.08)
  Pressing spontaneous pain LOCF endpoint (n=29,27) | 0.15 (0.06) | 0.08 (0.06)
  Paroxysmal pain Cycle 3 (n=27,24) | 0.00 (0.01) | 0.02 (0.01)
  Paroxysmal pain Cycle 4 (n=28,24) | 0.06 (0.06) | 0.13 (0.07)
  Paroxysmal pain Cycle 5 (n=25,24) | 0.06 (0.07) | 0.017 (0.07)
  Paroxysmal pain Cycle 6 (n=22,23) | 0.08 (0.09) | 0.21 (0.09)
  Paroxysmal pain Cycle 7(n=19,23) | 0.36 (0.17) | 0.35 (0.16)
  Paroxysmal pain Cycle 8 (n=18,21) | 0.63 (0.25) | 0.32 (0.23)
  Paroxysmal pain Cycle 9 (n=18,20) | 0.18 (0.17) | 0.38 (0.16)
  Paroxysmal pain LOCF endpoint (n=28,27) | 0.11 (0.10) | 0.20 (0.11)
  Evoke pain Cycle 2 (n=28,27) | 0.04 (0.06) | 0.04 (0.06)
  Evoke pain Cycle 3 (n=28,23) | 0.17 (0.11) | 0.07 (0.13)
  Evoke pain Cycle 4 (n=28,24) | 0.15 (0.08) | 0.28 (0.09)
  Evoke pain Cycle 5 (n=26,24) | 0.18 (0.14) | 0.29 (0.14)
  Evoke pain Cycle 6 (n=24,24) | 0.49 (0.28) | 0.66 (0.28)
  Evoke pain Cycle 7 (n=21,22) | 0.99 (0.26) | 0.40 (0.26)
  Evoke pain Cycle 8 (n=19,20) | 1.05 (0.36) | 0.36 (0.35)
  Evoke pain Cycle 9 (n=19,20) | 0.74 (0.26) | 0.59 (0.26)
  Evoke pain LOCF endpoint (n=29,27) | 0.46 (0.18) | 0.43 (0.19)
  Paresthesia/dysesthesia pain Cycle 2 (n=28,27) | 9.25 (0.08) | -0.00 (0.09)
  Paresthesia/dysesthesia pain Cycle 3(n=28,23) | 0.34 (0.10) | 0.14 (0.11)
  Paresthesia/dysesthesia pain Cycle 4 (n=28,24) | 0.43 (0.11) | 0.06 (0.12)
  Paresthesia/dysesthesia pain Cycle 5(n=26,24) | 0.60 (0.15) | 0.20 (0.15)
  Paresthesia/dysesthesia pain Cycle 6 (n=24,23) | 0.68 (0.23) | 0.32 (0.24)
  Paresthesia/dysesthesia pain Cycle 7 (n=21,22) | 0.78 (0.23) | 0.48 (0.22)
  Paresthesia/dysesthesia pain Cycle 8 (n=19,21) | 1.09 (0.34) | 0.58 (0.32)
  Paresthesia/dyesthesia pain Cycle 9 (n=18,20) | 1.17 (0.36) | 0.85 (0.34)
  Paresthesia/dyesthesia pain LOCF endpt (n=29,27) | 0.83 (0.24) | 0.52 (0.25)
  Total Score Cycle 2 (n=27,27) | 0.00 (0.00) | 0.00 (0.00)
  Total Score Cycle 3 (n=27,24) | 0.01 (0.00) | 0.00 (0.00)
  Total Score Cycle 4(n=27,23) | 0.01 (0.00) | 0.01 (0.00)
  Total Score Cycle 5 (n=25,24) | 0.01 (0.00) | 0.01 (0.00)
  Total Score Cycle 6(n=22,23) | 0.02 (0.01) | 0.02 (0.01)
  Total Score Cycle 7 (n=18,23) | 0.03 (0.02) | 0.02 (0.01)
  Total Score Cycle 8(n=18,20) | 0.04 (0.01) | 0.02 (0.01)
  Total Score Cycle 9 (n=17,20) | 0.03 (0.01) | 0.03 (0.01)
  Total Score Cycle LOCF Endpoint (n=28,27) | 0.02 (0.01) | 0.02 (0.01)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Burning Spontaneous Pain Cycle 3; Test type: Superiority or Other; p = 0.2034, ANCOVA; Mean Difference (Final Values) = 0.11, 95% CI [-0.06 to 0.29], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Burning Spontaneous Pain Cycle 4; Test type: Superiority or Other; p = 0.3062, ANCOVA; Mean Difference (Final Values) = -0.14, 95% CI [-0.40 to 0.13], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Burning Spontaneous Pain Cycle 5; Test type: Superiority or Other; p = 0.2787, ANCOVA; Mean Difference (Final Values) = -0.13, 95% CI [-0.37 to 0.11], Standard Error of Mean 0.12
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Burning Spontaneous Pain Cycle 6; Test type: Superiority or Other; p = 0.4124, ANCOVA; Mean Difference (Final Values) = 0.14, 95% CI [-0.20 to 0.47], Standard Error of Mean 0.17
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Burning Spontaneous Pain Cycle 7; Test type: Superiority or Other; p = 0.9541, ANCOVA; Mean Difference (Final Values) = 0.02, 95% CI [-0.68 to 0.73], Standard Error of Mean 0.35
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Burning Spontaneous Pain Cycle 8; Test type: Superiority or Other; p = 0.3383, ANOVA; Mean Difference (Final Values) = 0.30, 95% CI [-0.33 to 0.92], Standard Error of Mean 0.31
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Burning Spontaneous Pain; Test type: Superiority or Other; p = 0.8918, ANCOVA; Mean Difference (Final Values) = -0.05, 95% CI [-0.84 to 0.74], Standard Error of Mean 0.39
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Burning Spontaneous Pain LOCF endpoint; Test type: Superiority or Other; p = 0.9614, ANCOVA; Mean Difference (Final Values) = -0.01, 95% CI [-0.54 to 0.51], Standard Error of Mean 0.26
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Pressing Spontaneous Pain Cycle 2; Test type: Superiority or Other; p = 0.3022, ANCOVA; Mean Difference (Final Values) = -0.06, 95% CI [-0.17 to 0.05], Standard Error of Mean 0.06
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Pressing Spontaneous Pain Cycle 3; Test type: Superiority or Other; p = 0.3747, ANCOVA; Mean Difference (Final Values) = 0.04, 95% CI [-0.04 to 0.12], Standard Error of Mean 0.04
Statistical Analysis 11: Comparison: Pregabalin vs Placebo; Pressing Spontaneous Pain Cycle 4; Test type: Superiority or Other; p = 0.1630, ANCOVA; Mean Difference (Final Values) = -0.17, 95% CI [-0.40 to 0.07], Standard Error of Mean 0.12
Statistical Analysis 12: Comparison: Pregabalin vs Placebo; Pressing Spontaneous Pain Cycle 5; Test type: Superiority or Other; p = 0.9568, ANOVA; Mean Difference (Final Values) = -0.00, 95% CI [-0.12 to 0.11], Standard Error of Mean 0.06
Statistical Analysis 13: Comparison: Pregabalin vs Placebo; Pressing Spontaneous Pain Cycle 6; Test type: Superiority or Other; p = 0.9793, ANCOVA; Mean Difference (Final Values) = -0.00, 95% CI [-0.13 to 0.13], Standard Error of Mean 0.07
Statistical Analysis 14: Comparison: Pregabalin vs Placebo; Pressing Spontaneous Pain Cycle 7; Test type: Superiority or Other; p = 0.8850, ANCOVA; Mean Difference (Final Values) = -0.04, 95% CI [-0.54 to 0.47], Standard Deviation 0.25
Statistical Analysis 15: Comparison: Pregabalin vs Placebo; Pressing Spontaneous Pain Cycle 8; Test type: Superiority or Other; p = 0.2199, ANCOVA; Mean Difference (Final Values) = 0.27, 95% CI [-0.17 to 0.70], Standard Error of Mean 0.21
Statistical Analysis 16: Comparison: Pregabalin vs Placebo; Pressing Spontaneous Pain Cycle 9; Test type: Superiority or Other; p = 0.4017, ANCOVA; Mean Difference (Final Values) = 0.10, 95% CI [-0.14 to 0.35], Standard Error of Mean 0.12
Statistical Analysis 17: Comparison: Pregabalin vs Placebo; Pressing Spontaneous Pain LOCF Endpoint; Test type: Superiority or Other; p = 0.4113, ANCOVA; Mean Difference (Final Values) = 0.07, 95% CI [-0.10 to 0.24], Standard Error of Mean 0.09
Statistical Analysis 18: Comparison: Pregabalin vs Placebo; Paroxysmal Pain Cycle 3; Test type: Superiority or Other; p = 0.3011, ANCOVA; Mean Difference (Final Values) = -0.02, 95% CI [-0.06 to 0.02], Standard Error of Mean 0.02
Statistical Analysis 19: Comparison: Pregabalin vs Placebo; Paroxysmal Pain Cycle 4; Test type: Superiority or Other; p = 0.4482, ANCOVA; Mean Difference (Final Values) = -0.07, 95% CI [-0.26 to 0.12], Standard Error of Mean 0.10
Statistical Analysis 20: Comparison: Pregabalin vs Placebo; Paroxysmal Pain Cycle 5; Test type: Superiority or Other; p = 0.3058, ANCOVA; Mean Difference (Final Values) = -0.11, 95% CI [-0.31 to 0.10], Standard Error of Mean 0.10
Statistical Analysis 21: Comparison: Pregabalin vs Placebo; Paroxysmal Pain Cycle 6; Test type: Superiority or Other; p = 0.3035, ANCOVA; Mean Difference (Final Values) = -0.13, 95% CI [-0.38 to 0.12], Standard Error of Mean 0.12
Statistical Analysis 22: Comparison: Pregabalin vs Placebo; Paroxysmal Pain Cycle 7; Test type: Superiority or Other; p = 0.9636, ANCOVA; Mean Difference (Final Values) = 0.01, 95% CI [-0.46 to 0.48], Standard Error of Mean 0.23
Statistical Analysis 23: Comparison: Pregabalin vs Placebo; Paroxysmal Pain Cycle 8; Test type: Superiority or Other; p = 0.3660, ANCOVA; Mean Difference (Final Values) = 0.32, 95% CI [-0.38 to 1.02], Standard Error of Mean 0.35
Statistical Analysis 24: Comparison: Pregabalin vs Placebo; Paroxysmal Pain Cycle 9; Test type: Superiority or Other; p = 0.4093, ANCOVA; Mean Difference (Final Values) = -0.20, 95% CI [-0.69 to 0.29], Standard Error of Mean 0.24
Statistical Analysis 25: Comparison: Pregabalin vs Placebo; Paroxysmal Pain LOCF Endpoint; Test type: Superiority or Other; p = 0.5208, ANCOVA; Mean Difference (Final Values) = -0.10, 95% CI [-0.39 to 0.20], Standard Error of Mean 0.15
Statistical Analysis 26: Comparison: Pregabalin vs Placebo; Evoke Pain Cycle 2; Test type: Superiority or Other; p = 0.9931, ANCOVA; Mean Difference (Final Values) = 0.00, 95% CI [-0.17 to 0.17], Standard Error of Mean 0.08
Statistical Analysis 27: Comparison: Pregabalin vs Placebo; Evoke Pain Cycle 3; Test type: Superiority or Other; p = 0.5867, ANCOVA; Mean Difference (Final Values) = 0.09, 95% CI [-0.25 to 0.44], Standard Error of Mean 0.17
Statistical Analysis 28: Comparison: Pregabalin vs Placebo; Evoke Pain Cycle 4; Test type: Superiority or Other; p = 0.2748, ANCOVA; Mean Difference (Final Values) = -0.13, 95% CI [-0.37 to 0.11], Standard Error of Mean 0.12
Statistical Analysis 29: Comparison: Pregabalin vs Placebo; Evoke Pain Cycle 5; Test type: Superiority or Other; p = 0.5521, ANCOVA; Mean Difference (Final Values) = -0.12, 95% CI [-0.51 to 0.28], Standard Error of Mean 0.20
Statistical Analysis 30: Comparison: Pregabalin vs Placebo; Evoke Pain Cycle 6; Test type: Superiority or Other; p = 0.6734, ANCOVA; Mean Difference (Final Values) = -0.17, 95% CI [-0.96 to 0.62], Standard Error of Mean 0.39
Statistical Analysis 31: Comparison: Pregabalin vs Placebo; Evoke Pain Cycle 7; Test type: Superiority or Other; p = 0.1214, ANCOVA; Mean Difference (Final Values) = 0.58, 95% CI [-0.16 to 1.33], Standard Error of Mean 0.37
Statistical Analysis 32: Comparison: Pregabalin vs Placebo; Evoke Pain Cycle 8; Test type: Superiority or Other; p = 0.1845, ANCOVA; Mean Difference (Final Values) = 0.69, 95% CI [-0.34 to 1.72], Standard Error of Mean 0.51
Statistical Analysis 33: Comparison: Pregabalin vs Placebo; Evoke Pain Cycle 9; Test type: Superiority or Other; p = 0.6863, ANCOVA; Mean Difference (Final Values) = 0.15, 95% CI [-0.60 to 0.90], Standard Error of Mean 0.37
Statistical Analysis 34: Comparison: Pregabalin vs Placebo; Evoke Pain LOCF Endpoint; Test type: Superiority or Other; p = 0.9273, ANCOVA; Mean Difference (Final Values) = 0.02, 95% CI [-0.51 to 0.56], Standard Error of Mean 0.27
Statistical Analysis 35: Comparison: Pregabalin vs Placebo; Parethesia/Dysesthesia Pain Cycle 2; Test type: Superiority or Other; p = 0.0416, ANCOVA; Mean Difference (Final Values) = 0.25, 95% CI [0.01 to 0.50], Standard Error of Mean 0.12
Statistical Analysis 36: Comparison: Pregabalin vs Placebo; Parethesia/Dysesthesia Pain Cycle 3; Test type: Superiority or Other; p = 0.1819, ANCOVA; Mean Difference (Final Values) = 0.20, 95% CI [-0.10 to 0.50], Standard Error of Mean 0.15
Statistical Analysis 37: Comparison: Pregabalin vs Placebo; Parethesia/Dysesthesia Pain Cycle 4; Test type: Superiority or Other; p = 0.0331, ANCOVA; Mean Difference (Final Values) = 0.37, 95% CI [0.03 to 0.70], Standard Error of Mean 0.17
Statistical Analysis 38: Comparison: Pregabalin vs Placebo; Parethesia/Dysesthesia Pain Cycle 5; Test type: Superiority or Other; p = 0.0608, ANCOVA; Mean Difference (Final Values) = 0.40, 95% CI [-0.02 to 0.83], Standard Error of Mean 0.21
Statistical Analysis 39: Comparison: Pregabalin vs Placebo; Parethesia/Dysesthesia Pain Cycle 6; Test type: Superiority or Other; p = 0.2809, ANCOVA; Mean Difference (Final Values) = 0.36, 95% CI [-0.31 to 1.03], Standard Error of Mean 0.33
Statistical Analysis 40: Comparison: Pregabalin vs Placebo; Parethesia/Dysesthesia Pain Cycle 7; Test type: Superiority or Other; p = 0.3445, ANCOVA; Mean Difference (Final Values) = 0.31, 95% CI [-0.34 to 0.95], Standard Error of Mean 0.32
Statistical Analysis 41: Comparison: Pregabalin vs Placebo; Parethesia/Dysesthesia Pain Cycle 8; Test type: Superiority or Other; p = 0.2806, ANCOVA; Mean Difference (Final Values) = 0.51, 95% CI [-0.44 to 1.46], Standard Error of Mean 0.47
Statistical Analysis 42: Comparison: Pregabalin vs Placebo; Parethesia/Dysesthesia Pain Cycle 9; Test type: Superiority or Other; p = 0.5217, ANCOVA; Mean Difference (Final Values) = 0.32, 95% CI [-0.68 to 1.33], Standard Error of Mean 0.49
Statistical Analysis 43: Comparison: Pregabalin vs Placebo; Parethesia/Dysesthesia Pain LOCF Endpoint; Test type: Superiority or Other; p = 0.3628, ANCOVA; Mean Difference (Final Values) = 0.31, 95% CI [-0.37 to 1.00], Standard Error of Mean 0.34
Statistical Analysis 44: Comparison: Pregabalin vs Placebo; Total Score Cycle 2; Test type: Superiority or Other; p = 0.3557, ANCOVA; Mean Difference (Final Values) = 0.00, 95% CI [-0.00 to 0.01], Standard Error of Mean 0.00
Statistical Analysis 45: Comparison: Pregabalin vs Placebo; Total Score Cycle 3; Test type: Superiority or Other; p = 0.2824, ANCOVA; Mean Difference (Final Values) = 0.00, 95% CI [-0.00 to 0.01], Standard Error of Mean 0.00
Statistical Analysis 46: Comparison: Pregabalin vs Placebo; Total Score Cycle 4; Test type: Superiority or Other; p = 0.5931, ANCOVA; Mean Difference (Final Values) = -0.00, 95% CI [-0.01 to 0.01], Standard Error of Mean 0.00
Statistical Analysis 47: Comparison: Pregabalin vs Placebo; Total Score Cycle 5; Test type: Superiority or Other; p = 0.9865, ANCOVA; Mean Difference (Final Values) = -0.00, 95% CI [-0.01 to 0.01], Standard Error of Mean 0.00
Statistical Analysis 48: Comparison: Pregabalin vs Placebo; Total Score Cycle 6; Test type: Superiority or Other; p = 0.9854, ANCOVA; Mean Difference (Final Values) = -0.00, 95% CI [-0.02 to 0.02], Standard Error of Mean 0.01
Statistical Analysis 49: Comparison: Pregabalin vs Placebo; Total Score Cycle 7; Test type: Superiority or Other; p = 0.3403, ANCOVA; Mean Difference (Final Values) = 0.01, 95% CI [-0.01 to 0.04], Standard Error of Mean 0.01
Statistical Analysis 50: Comparison: Pregabalin vs Placebo; Total Score Cycle 8; Test type: Superiority or Other; p = 0.2226, ANCOVA; Mean Difference (Final Values) = 0.02, 95% CI [-0.01 to 0.05], Standard Error of Mean 0.02
Statistical Analysis 51: Comparison: Pregabalin vs Placebo; Total Score Cycle 9; Test type: Superiority or Other; p = 0.9694, ANCOVA; Mean Difference (Final Values) = 0.00, 95% CI [-0.03 to 0.03], Standard Error of Mean 0.01
Statistical Analysis 52: Comparison: Pregabalin vs Placebo; Total Score LOCF Endpoint; Test type: Superiority or Other; p = 0.8957, ANCOVA; Mean Difference (Final Values) = 0.00, 95% CI [-0.02 to 0.02], Standard Error of Mean 0.01

5. Secondary Outcome: Number of Participants With Persistent Paresthesic, Dysesthesic, and Pain Symptoms
Description: Number of participants with persistent paresthesic, dyesthesic, and pain symptoms at chemotherapy Cycle 9 and last observation carried forward (LOCF) endpoint. Numeric rating scale of symptoms: >=1: mild symptoms to >=4: moderate severe symptoms. Subjects rated their average severity of symptoms over the last 24 hours every evening before bedtime.
Time Frame: Cycle 9 and Last Observation Carried Forward (LOCF) cycle endpoint
Population: ITT population, subjects with at least 1 dose of study medication and for whom at least 1 post-baseline efficacy evaluation was obtained.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 32 | 29
participants
  Paresthesia Cycle 9 (n=19,19) (>or=1) | 7 | 6
  Paresthesia LOCF endpoint (n=30,29) (>or=1) | 8 | 7
  Paresthesia Cycle 9 (n=19,19) (>or=2) | 4 | 3
  Paresthesia LOCF endpoint (n=30,29) (>or=2) | 5 | 3
  Paresthesia Cycle 9 (n=19,19) (>or=3) | 2 | 1
  Paresthesia LOCF endpoint (n=30,29) (>or=3) | 3 | 1
  Paresthesia Cycle 9 (n=19,19) (>or=4) | 1 | 1
  Paresthesia LOCF endpoint (n=30,29) (>or=4) | 2 | 1
  Dysesthesia Cycle 9 (n=19,19) (>or=1) | 10 | 4
  Dysesthesia LOCF endpoint (n=30,29) (>or=1) | 11 | 5
  Dysesthesia Cycle 9 (n=19,19) (>or=2) | 5 | 3
  Dysesthesia LOCF endpoint (n=30,29) (>or=2) | 6 | 4
  Dysesthesia Cycle 9 (n=19,19) (>or=3) | 3 | 1
  Dysesthesia LOCF endpoint (n=30,29) (>or=3) | 4 | 2
  Dysesthesia Cycle 9 (n=19,19) (>or=4) | 1 | 1
  Dysesthesia LOCF endpoint (n=30,29 (>or=4) | 2 | 2
  Pain Cycle 9 (n=19,19) (>or=1) | 6 | 2
  Pain LOCF endpoint (n=30,29;) (>or=1) | 6 | 3
  Pain Cycle 9 (n=19,19) (>or=2) | 2 | 1
  Pain LOCF endpoint (n=30,29) (>or=2) | 2 | 2
  Pain Cycle 9 (n=19,19) (>or=3) | 1 | 1
  Pain LOCF endpoint (n=30,29) (>or=3) | 1 | 2
  Pain Cycle 9 (n=19,19) (>or=4) | 0 | 1
  Pain LOCF endpoint (n=30,29) (>or=4) | 0 | 2

6. Primary Outcome: Duration Adjusted Average Change (DAAC) of Paresthesia From the Onset of Chemotherapy Measured by Numeric Rating Scale (NRS)
Description: Least squares mean of change: mean at cycle minus mean at Baseline. Paresthetic duration Adjusted Average Change (DAAC) endpoint was computed based on Numeric Rating Scale (NRS) of paresthesia (collected 0=no pain; 1-3=mild pain; 4-6=moderate pain; 7-10=severe pain). DAAC endpoint is defined as the Area Under Curve (AUC) of the collected NRS over time, divided by the collection time period (up to 10 days).
Time Frame: Period of 10 days from the onset of chemotherapy to the last cycle: Last Observation Carried Forward (LOCF)
Population: Intent-to-Treat (ITT) population: subjects with at least 1 dose of study medication and for whom at least 1 post-baseline efficacy evaluation was obtained; Last Observation Carried Forward (LOCF): last recorded cycle. Primary analysis timeframe: 10 days of paresthesia scores from the onset of chemotherapy to the last cycle of chemotherapy (LOCF).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 32 | 29
score on scale | 1.11 (0.35) | 1.27 (0.34)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; LOCF cycle endpoint. Sample size based on original primary efficacy parameter (PEP) of time to persistent symptoms (developing in 35% of pregabalin subjects & 60% of placebo subjects). Assuming Type I error rate of 0.05 and a 2-sided log-rank test for equality of time to persistent symptoms survival curves, study would have had at least 90% power using 100 subjects per treatment group. Original PEP was modified to secondary due to lack of persistent paresthetic symptom emergence; Test type: Superiority or Other; p = 0.7489, ANCOVA — No multiple comparisons adjustment was necessary; Model terms include treatment, study center, and baseline score; Median Difference (Final Values) = -0.16, Standard Error of Mean 0.49 — Least squares (LS) means and corresponding standard errors derived from ANCOVA model were used

ADVERSE EVENTS:
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 5/32 | 7/29
Other Adverse Events (participants affected / at risk) | 31/32 | 27/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=32) | Placebo (N=29)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Vitreous hemorrhage (Eye disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Disease progression (General disorders) | 0 | 1
Extravasation (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Peritoneal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Shock (Vascular disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=32) | Placebo (N=29)
Neutropenia (Blood and lymphatic system disorders) | 9 | 10
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Leukopenia (Blood and lymphatic system disorders) | 5 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 8
Tachycardia (Cardiac disorders) | 0 | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Eye irritation (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 5
Constipation (Gastrointestinal disorders) | 8 | 8
Diarrhoea (Gastrointestinal disorders) | 9 | 8
Dry mouth (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 2
Gingival pain (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 16 | 13
Oesophageal pain (Gastrointestinal disorders) | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0
Rectal tenesmus (Gastrointestinal disorders) | 1 | 1
Stomatitis (Eye disorders) | 3 | 5
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 5 | 10
Asthenia (General disorders) | 7 | 4
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 4 | 2
Fatigue (General disorders) | 8 | 7
Feeling cold (General disorders) | 1 | 1
Implant site pain (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 6 | 5
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Peripheral coldness (General disorders) | 0 | 2
Pyrexia (General disorders) | 8 | 4
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 2
Allergy to arthropod sting (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 3
Hypersensitivity (Immune system disorders) | 1 | 1
Cystitis (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 4
Otitis media (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatine increased (Investigations) | 1 | 0
Body temperature increased (Investigations) | 1 | 0
Platelet count (Investigations) | 1 | 1
Weight decreased (Investigations) | 1 | 1
Weight increased (Investigations) | 0 | 3
Anorexia (Metabolism and nutrition disorders) | 13 | 11
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Neckpain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Amnesia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 7 | 4
Dysaethesia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 5 | 2
Hyperaesthesia (Nervous system disorders) | 1 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 7 | 7
Paraesthesia (Nervous system disorders) | 1 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 3
Polyneuropathy (Nervous system disorders) | 0 | 2
Syncope vasovagal (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 5
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Balanitis (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 4
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 4
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2
Circulatory collapse (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 2 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
hypoaesthesia (Nervous system disorders) | 2 | 2

LIMITATIONS AND CAVEATS:
Due to lack of symptom emergence, enrollment was halted, and endpoint modified because primary assumptions upon which it was powered (emergence of symptomatology) were not met, and not all endpoints were able to be reliably analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.